CLINICAL TRIAL: NCT02730689
Title: A Randomized, Single-dose, Open, Crossover Clinical Trial to Compare the Pharmacokinetics of DP-R207 in Comparison to Each Component Administered Alone in Healthy Male Volunteers
Brief Title: A Study to Compare the Pharmacokinetics of DP-R207 in Comparison to Each Component Administered Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DP-CTR207-I-03
Record Dates: First submitted 2016-03-16; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Volunteers
Keywords: DP-R207; Rosuvastatin; Ezetimibe
MeSH Terms: interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A group (Experimental): DP-R207 >> rosuvastatin+ezetimibe
  Interventions: Drug: DP-R207; Drug: Rosuvastatin; Drug: Ezetimibe
- B group (Active Comparator): rosuvastatin+ezetimibe >> DP-R207
  Interventions: Drug: DP-R207; Drug: Rosuvastatin; Drug: Ezetimibe

INTERVENTIONS:
Drug: DP-R207
Drug: Rosuvastatin
Drug: Ezetimibe

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of DP-R207 (Rosuvastatin 10mg and Ezetimibe 10mg fixed dose combinations) in comparison to each component administered alone in health male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects age between 19 and 55 signed informed consent

Exclusion Criteria:

* subjects have an allergy reaction of this drug

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 0-72hr
Peak Plasma Concentration (Cmax) | 0-72hr